CLINICAL TRIAL: NCT01267552
Title: Randomized Clinical Trial of Axillary Lymphadenectomy Without Drainage for Breast Cancer Treatment
Brief Title: Study of Axillary Lymphadenectomy Without Drainage for Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Araujo Jorge Hospital (Other)
Responsible Party: Ruffo Freitas-Junior, Federal University of Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Drains Trial; Drains trial01/2007 (Registry Identifier: FAPEG 01/2007)
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer; Complications; Seroma
Keywords: Breast cancer; Surgery; Complications; Drainage; Seroma
MeSH Terms: conditions — Breast Neoplasms; Seroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non drainage arm (Experimental): No drains will be placed during operation
  Interventions: Procedure: Non drains will be placed during operation
- Drainage arm (Active Comparator): Closed suction drains will be placed during operation
  Interventions: Procedure: Closed suction drainage

INTERVENTIONS:
Procedure: Non drains will be placed during operation — Non drains will be placed during operation
  Other Names: No drainage
  Arms: Non drainage arm
Procedure: Closed suction drainage — Closed suction drainage will be placed during operation
  Arms: Drainage arm

SUMMARY:
To study the safety of not draining the axilla, after breast conserving surgery and full axillary lymphadenectomy.

DETAILED DESCRIPTION:
The primary objective is to study the safety of not draining the axilla, considering the total number of patients without complication among breast cancer patients treated by means of conservative surgery and full axillary lymphadenectomy, with or without axillary drainage.

The secondary objectives will be the numbers of aspiration punctures, volumes of fluid aspirated and the total volumes of fluid produced.

ELIGIBILITY:
Inclusion Criteria:

* Stage I and II breast cancer patients
* Will be submitted to breast conserving therapy, with full axillary lymphadenectomy

Exclusion Criteria:

* diabetes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2000-07; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  The safety of not draining the axilla, will be considered by the total number of patients without complication among breast cancer patients treated by means of breast conserving surgery and full axillary lymphadenectomy

SECONDARY OUTCOMES:
Serous fluid | 6 months
  The number of aspiration punctures; Volume of fluid aspirated; Total volumes of fluid produced

CONTACTS AND LOCATIONS:
Overall Officials: Ruffo Freitas-Junior, PhD, Principal Investigator — Universidade Federal de Goias; Luiz Fernando J Ribeiro, PhD, Study Chair — Hospital Araujo Jorge, Associacao de Combate ao Cancer em Goias
Locations (2):
- Brazil (2):
  - Hospital Araujo Jorge, Associacao de Combate ao Cancer em Goias, Goiânia, Goiás
  - Mastology Program of Federal University of Goias, Goiânia, Goiás

REFERENCES:
- [Derived] Freitas-Junior R, Ribeiro LFJ, Moreira MAR, Queiroz GS, Esperidiao MD, Silva MAC, Pereira RJ, Zampronha RAC, Rahal RMS, Soares LR, Dos Santos DL, Thomazini MV, de Faria CFS, Paulinelli RR. Complete axillary dissection without drainage for the surgical treatment of breast cancer: a randomized clinical trial. Clinics (Sao Paulo). 2017 Jul;72(7):426-431. doi: 10.6061/clinics/2017(07)07. PMID 28793003